CLINICAL TRIAL: NCT00958906
Title: Pilot Study for the Evaluation of Intravitreal Infliximab in the Treatment of Uveitic Macular Edema
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left institution (there are no data results for this study)
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Farzin Forooghian, MD, Assistant Professor, Department of Ophthalmology, Mount Sinai School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO # 09-0611
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Uveitic Macular Edema; Intraocular Inflammation
Keywords: Infliximab; Uveitis; Macular Edema; Intraocular Inflammation
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal infliximab (Experimental)
  Interventions: Drug: Infliximab (intravitreal, 2.0mg/0.05ml)

INTERVENTIONS:
Drug: Infliximab (intravitreal, 2.0mg/0.05ml) — One injection of intravitreal infliximab (2.0mg/0.05ml).
  Other Names: Remicade™

SUMMARY:
The purpose of this study is to determine if intravitreal infliximab is a safe and effective treatment for macular edema secondary to uveitis.

DETAILED DESCRIPTION:
Participants with uveitic macular edema will be treated with one injection of intravitreal infliximab (2.0mg/0.05ml) and followed for three months. Outcomes that be assessed include best-corrected visual acuity, macular thickness as measured by optical coherence tomography, and electroretinogram responses.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Participants must have uveitic macular edema in one eye as defined by all of the following criteria:

   1. Presence of active intermediate uveitis or posterior uveitis.
   2. Macular edema defined as a central macular thickness of ≥ 250 μm on OCT.
   3. Uveitis must be noninfectious as determined by standard investigations used in the diagnostic investigation of uveitis.
4. Participant must have visual acuity between 20/40 and hand motions in the study eye.
5. Participant must have a steady fixation in the study eye and media clear enough for good quality imaging.
6. Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must practice an adequate method of birth control. Males able to father a child must agree to practice birth control. Acceptable methods of birth control include hormonal contraception (birth control pills, injected hormones or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom and spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy in a partner). If a participant is of childbearing potential, she must be willing to undergo monthly urine pregnancy tests. Both males and females must agree to use adequate birth control for three months after the intravitreal infliximab injection.

Exclusion Criteria:

1. Participant is in another investigational study and actively receiving study therapy.
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant has uveitic macular edema (as defined above) in both eyes.
4. Participant has multiple sclerosis or symptoms suggestive of multiple sclerosis.
5. Participant has evidence of ocular disease other than uveitis in either eye that may confound the outcome of the study (e.g., diabetic retinopathy, age-related macular degeneration, vitreomacular traction, moderate/severe myopia, etc.).
6. Participant is expected to need ocular surgery in the study eye during the course of the study.
7. Participant has undergone ocular surgery or an intravitreal/periocular steroid injection in the study eye within the past 3 months.
8. Participant has had a YAG laser capsulotomy or intravitreal anti-VEGF treatment in the study eye within the past 6 weeks.
9. Participant has had a pars plana vitrectomy in the study eye.
10. Participant is on ocular or systemic medications known to be toxic to the lens, retina, or optic nerve.
11. Participant with a history of ocular herpes simplex virus infection in the study eye.
12. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
13. There are no criteria for inclusion/exclusion for the fellow eye. Only one eye can have macular edema in order for the potential participant to be considered for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-08; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | Three months

SECONDARY OUTCOMES:
Macular thickness | One, two, and three months

CONTACTS AND LOCATIONS:
Overall Officials: Farzin Forooghian, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Department of Ophthalmology, Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Theodossiadis PG, Liarakos VS, Sfikakis PP, Vergados IA, Theodossiadis GP. Intravitreal administration of the anti-tumor necrosis factor agent infliximab for neovascular age-related macular degeneration. Am J Ophthalmol. 2009 May;147(5):825-30, 830.e1. doi: 10.1016/j.ajo.2008.12.004. Epub 2009 Feb 10. PMID 19211094
- [Background] Theodossiadis PG, Liarakos VS, Sfikakis PP, Charonis A, Agrogiannis G, Kavantzas N, Vergados IA. Intravitreal administration of the anti-TNF monoclonal antibody infliximab in the rabbit. Graefes Arch Clin Exp Ophthalmol. 2009 Feb;247(2):273-81. doi: 10.1007/s00417-008-0967-4. Epub 2008 Nov 4. PMID 18982345
- [Background] Giansanti F, Ramazzotti M, Vannozzi L, Rapizzi E, Fiore T, Iaccheri B, Degl' Innocenti D, Moncini D, Menchini U. A pilot study on ocular safety of intravitreal infliximab in a rabbit model. Invest Ophthalmol Vis Sci. 2008 Mar;49(3):1151-6. doi: 10.1167/iovs.07-0932. PMID 18326743
- [Background] Olson JL, Courtney RJ, Mandava N. Intravitreal infliximab and choroidal neovascularization in an animal model. Arch Ophthalmol. 2007 Sep;125(9):1221-4. doi: 10.1001/archopht.125.9.1221. PMID 17846362